CLINICAL TRIAL: NCT00887406
Title: A Study to Evaluate the Safety, Tolerability, Systemic Pharmacokinetic Profile and Pharmacodynamics of Single and Repeat Inhaled Doses of GSK961081 in Healthy Subjects
Brief Title: Study of GSK961081 in Healthy Volunteer Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Theravance Biopharma (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 104865
Record Dates: First submitted 2009-04-23; First posted 2009-04-24 (Estimated); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: first time in human study; COPD; long-acting bronchodilator
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — batefenterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (10):
- Cohort 1, Period 2 (Experimental): GSK961081 3mcg, Placebo, GSK961081 15mcg, GSK961081 50mcg
  Interventions: Drug: GSK961081 15mcg SD; Drug: GSK961081 3mcg SD; Drug: GSK961081 50mcg SD; Drug: Placebo SD
- Cohort 1, period 1 (Experimental): Placebo, GSK961081 3mcg, GSK961081 15mcg, GSK961081 50mcg
  Interventions: Drug: GSK961081 15mcg SD; Drug: GSK961081 3mcg SD; Drug: GSK961081 50mcg SD; Drug: Placebo SD
- Cohort 1, period 3 (Experimental): GSK961081 3mcg, GSK961081 15mcg, Placebo, GSK961081 50mcg
  Interventions: Drug: GSK961081 15mcg SD; Drug: GSK961081 3mcg SD; Drug: GSK961081 50mcg SD; Drug: Placebo SD
- Cohort 1, period 4 (Experimental): GSK961081 3mcg, GSK961081 15mcg, GSK961081 50mcg, Placebo
  Interventions: Drug: GSK961081 15mcg SD; Drug: GSK961081 3mcg SD; Drug: GSK961081 50mcg SD; Drug: Placebo SD
- Cohort 2, period 1 (Experimental): Placebo, GSK961081 100mcg, GSK961081 200mcg, GSK961081 300mcg,
  Interventions: Drug: Placebo SD; Drug: GSK961081 100mcg SD; Drug: GSK961081 200mcg SD; Drug: GSK961081 300mcg SD
- Cohort 2, period 2 (Experimental): GSK961081 100mcg, Placebo, GSK961081 200mcg, GSK961081 300mcg
  Interventions: Drug: Placebo SD; Drug: GSK961081 100mcg SD; Drug: GSK961081 200mcg SD; Drug: GSK961081 300mcg SD
- Cohort 2, period 3 (Experimental): GSK961081 100mcg, GSK961081 200mcg, Placebo, GSK961081 300mcg
  Interventions: Drug: Placebo SD; Drug: GSK961081 100mcg SD; Drug: GSK961081 200mcg SD; Drug: GSK961081 300mcg SD
- Cohort 2, period 4 (Experimental): GSK961081 100mcg, GSK961081 200mcg, GSK961081 300mcg, Placebo
  Interventions: Drug: Placebo SD; Drug: GSK961081 100mcg SD; Drug: GSK961081 200mcg SD; Drug: GSK961081 300mcg SD
- Cohort 3 (Experimental): GSK961081 100mcg or Placebo
  Interventions: Drug: GSK961081 100mcg RD; Drug: Placebo RD
- Cohort 4 (Experimental): GSK961081 300mcg or Placebo
  Interventions: Drug: GSK961081 300mcg RD; Drug: Placebo RD

INTERVENTIONS:
Drug: GSK961081 15mcg SD — Single dose delivered via solution for nebulisation
  Other Names: Placebo; GSK961081 200mcg SD; GSK961081 50mcg SD; GSK961081 300mcg SD; GSK961081 100mcg SD; GSK961081 3mcg SD
  Arms: Cohort 1, Period 2; Cohort 1, period 1; Cohort 1, period 3; Cohort 1, period 4
Drug: GSK961081 3mcg SD — single dose delivered via nebulsier
  Arms: Cohort 1, Period 2; Cohort 1, period 1; Cohort 1, period 3; Cohort 1, period 4
Drug: GSK961081 50mcg SD — single dose delivered via solution for nebulisation
  Arms: Cohort 1, Period 2; Cohort 1, period 1; Cohort 1, period 3; Cohort 1, period 4
Drug: Placebo SD — single dose via nebuliser
  Arms: Cohort 1, Period 2; Cohort 1, period 1; Cohort 1, period 3; Cohort 1, period 4; Cohort 2, period 1; Cohort 2, period 2; Cohort 2, period 3; Cohort 2, period 4
Drug: GSK961081 100mcg SD — single dose delivered via solution for nebulisation
  Arms: Cohort 2, period 1; Cohort 2, period 2; Cohort 2, period 3; Cohort 2, period 4
Drug: GSK961081 200mcg SD — single dose via nebuliser
  Arms: Cohort 2, period 1; Cohort 2, period 2; Cohort 2, period 3; Cohort 2, period 4
Drug: GSK961081 300mcg SD — single dose via nebuliser
  Arms: Cohort 2, period 1; Cohort 2, period 2; Cohort 2, period 3; Cohort 2, period 4
Drug: GSK961081 100mcg RD — repeat dose via nebuliser
  Other Names: GSK961081 100mcg SD
  Arms: Cohort 3
Drug: GSK961081 300mcg RD — repeat dose vai nebuliser
  Arms: Cohort 4
Drug: Placebo RD — repeat dose via nebuliser
  Arms: Cohort 3; Cohort 4

SUMMARY:
GSK961081 is a new long-acting bronchodilator being developed for the treatment of chronic obstructive pulmonary disease (COPD). This study is the first clinical study in humans. The purpose of this study is to determine the safety, tolerability, pharmacokinetics and pharmacodynamics of GSK961081 in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males aged between 18 and 50 years.
* Body mass index within the range 18.5-29.9 kilograms/meter2 (kg/m2).
* Forced Expiratory Volume in 1 second (FEV1) <80% predicted and a FEV1/ Forced Vital Capacity (FVC) ratio <0.7
* Response to Salbutamol defined as: an increase in sGAW of >15% over pre-dose baseline within 2 h following administration of 400 mcg Salbutamol by MDI inhaler OR: a documented increase in sGAW of >15% over pre-dose baseline within 2 h following administration of 400 mcg Salbutamol by MDI inhaler within 6 months of screening.
* Response to Ipratropium bromide defined as: an increase in sGaw of >25% over pre-dose baseline within 2 h following 80 mcg Ipratropium bromide; OR: a documented increase in sGaw of >25% over pre-dose baseline 2 h following administration of 80 mcg Ipratropium bromide within 6 months of screening.
* A signed and dated written informed consent is obtained for the subject
* The subject is able to understand and comply with the protocol requirements, instructions and protocol-stated restrictions.
* Subjects who are current non-smokers who have not used any tobacco products in the 6-month period preceding the screening visit and have a pack history of > or = 10 pack years.

[number of pack years = (number of cigarettes per day/20) x number of years smoked]

Exclusion Criteria:

* Any clinically relevant abnormality identified at the screening medical assessment (physical examination/medical history), clinical laboratory tests, or ECG (12-lead or Holter).
* A history of breathing problems (i.e. history of asthmatic symptoms). Screening lung function tests (FEV1, FVC and sGaw) will be performed to confirm normal lung function parameters.
* A mean QTc(B) and QTc(F) value at screening >430msec, the 3 screening ECGs are not within 10% of the mean, a PR interval outside the range 120-210msec or an ECG that is not suitable for QT measurements (e.g. poorly defined termination of the T wave).
* A supine blood pressure that is persistently higher than 140/90 millimetres of mercury (mmHg) at screening.
* A supine mean heart rate outside the range 40-90 beats per minute (bpm) at screening.
* The subject has donated a unit of blood within the 90 days or intends to donate within 90 days after completing the study.
* A history of claustrophobia such that they may not tolerate plethysmography measurements.
* The subject is currently taking regular (or course of) medication whether prescribed or not, including vitamins and herbal remedies such as St John's Wort.
* The subject has used prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (which ever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and Sponsor the medication will not interfere with the study procedures or compromise subject safety.
* The subject has participated in a clinical study with another New Chemical Entity (NCE) within the past 112 days or a clinical study with any other drug during the previous 84 days.
* The subject is infected with the Hepatitis B, Hepatitis C, or HIV virus.
* The subject has a positive pre-study urine cotinine/ breath carbon monoxide test, urine drug/urine alcohol screen. A minimum list of drugs that will be screened for include Amphetamines, Barbituates, Cocaine, Opiates, Cannabinoids and Benzodiazepines.
* A history of regular alcohol consumption exceeding weekly intake of alcohol greater than 28 units, or an average daily intake of greater than 4 units.
* Are unable to use the Prodose AAD nebuliser device correctly.
* An unwillingness of subjects to abstain from sexual intercourse with pregnant or lactating women; or an unwillingness of the subject to use a condom/spermicide in addition to having their female partner use another form of contraception such as IUD, diaphragm with spermicide, oral contraceptives, injectable progesterone, subdermal implants or tubal ligation if the woman could become pregnant from the time of the first dose study medication until 90 days post-dose.
* The subject has a history of drug or other allergy, which, in the opinion of the responsible physician, contraindicates their participation.
* The subject has a history of hypersensitivity to Salbutamol or Ipratropium bromide, and for those subjects in cohorts III and IV, hypersensitivity to a beta-blocker.
* The subject has had a lower respiratory tract infection within 4 weeks of study start

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2005-11-07 (Actual); Primary Completion 2006-10-04 (Actual); Study Completion 2006-10-04 (Actual)

PRIMARY OUTCOMES:
General safety and tolerability (adverse events, clinical laboratory safety tests, cardiac monitoring, vital signs (including postural changes in blood pressure), 12-lead ECG parameters including QTc(b) and QTc(f), blood glucose and serum potassium). | Pre and post-dose on Days 1, 4 and 7

SECONDARY OUTCOMES:
Maxiumum and weighted mean (over 0-8 hours post-dose) for systolic and diastolic blood pressure, heart rate, QTc(F), QTc(B), plasma glucose and serum potassium | Days 1, 4 and 7
specific airway conductance (sGaW) | pre and post-dose on Days 1, 4 and 7
forced expiratory volume in one second (FEV1) | Pre and post-dose on Days 1, 4 and 7

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 104865 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/104865?search=study&search_terms=104865#rs
- Available data/document: Individual Participant Data Set: 104865 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 104865 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 104865 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 104865 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 104865 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 104865 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register